CLINICAL TRIAL: NCT06638138
Title: A Multi-center, Prospective, Blinded, Randomized Study of Artelon FLEXBAND® for Patients Undergoing Soft Tissue Reconstruction of the Anterior Talofibular Ligament (ATFL) to Treat Lateral Ankle Instability
Brief Title: Study of Artelon FLEXBAND® for Patients Undergoing Soft Tissue Reconstruction of the Anterior Talofibular Ligament (ATFL) to Treat Lateral Ankle Instability
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ART-003
Record Dates: First submitted 2024-09-05; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Lateral Ankle Instability
Keywords: ATFL reconstructive procedure; Flexband; modified Bröstrom reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FLEXBAND (Active Comparator): This group will undergo a lateral ankle ligament repair using the modified Broström technique with Artelon FLEXBAND augmentation of the ATFL.
  Interventions: Device: Flexband
- Control (No Intervention): This group will undergo a lateral ankle ligament repair using the modified Broström technique. This technique utilizes anchors to repair the ATFL, in some cases the CFL, lateral ankle capsule and extensor retinaculum. This will be done without Artelon FLEXBAND augmentation.

INTERVENTIONS:
Device: Flexband — Artelon FLEXBAND is a commercially available, polycaprolactone polyurethane urea (PCL/PUUR) multipolymer synthetic knitted mesh that is used for soft tissue reinforcement procedures. The device is biocompatible and degradable and has been used as an augmentation device in over 50,000 Orthopedic tendon and ligament reconstructive procedures. The FLEXBAND kits contain the device and all of the instrumentation needed to insert the device.
  Arms: FLEXBAND

SUMMARY:
The goal of this clinical trial is to analzye return to pre-injury activity level on study participants with lateral ankle instability undergoing a modified Bröstrom reconstruction procedure for repair of the ATFL. Study participants undergoing ATFL reconstructive procedure using the ARTELON FLEXBAND System as an augmentation device will be compared to study participants undergoing a standard modified Bröstrom procedure alone. Clinician reported safety and functional outcomes measures will be collected at baseline; and at 2-, 6-, 12-, 18 and 26-weeks and 1- and 2-years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between and including the age of 18-75 at the time of surgery.
2. Subjects who were diagnosed with lateral ankle instability by physician clinical assessment.
3. Subjects who will undergo a modified Bröstrom procedure for an ATFL repair with or without FLEXBAND augmentation device (does not require an isolated repair).
4. Subjects that are able to understand, complete and sign the Consent Form.

Exclusion Criteria:

1. Significant secondary procedures done at the time of repair, including significant osteochondral lesions and/or significant microfracture of the talus or tibia that warrant modifying the typical lateral ligament repair post-op rehab protocol (minor microfractures and OCD lesions that do not warrant major bone debridement, synovectomies, and bone spur/osteophyte removals are allowed).
2. Any concomitant orthopedic procedure that will extend the post-op rehabilitation (e.g., casting/immobilization) beyond the routinely prescribed rehab protocol following an ATFL reconstructive procedure.
3. Subjects undergoing a Calcaneal osteotomy.
4. Subjects requiring major additional tendon surgery (i.e., peroneal tendon repair or tenodesis).
5. Neuropathy.
6. Subjects with diabetes, who, in the opinion of the investigator, are not sufficiently controlled.
7. BMI greater than 40 kg/m2.
8. Subjects with active Worker's Compensation Cases
9. Any subject with a history of infection of the ankle predating the ankle repair.
10. Subjects with a systemic ligament laxity disorder (i.e., Ehlers-Danlos Syndrome).
11. Any orthopedic issue outside of the ankle that the Investigator feels may impede functional endpoint outcome measures.
12. Subjects who have a medical history that would likely make the subject an unreliable research participant.
13. Subjects that are nursing or pregnant at the time of surgery.
14. Subjects with physician assessed untreated alcohol or substance abuse at the time of screening.
15. Subjects who are currently enrolled or participated in another investigational device, drug, or biological trial within 60 days of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2027-06-23 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | From 2 weeks post-surgery to 26 weeks post-surgery.
  The primary outcome measure will be subject reported assessment of time to pre-injury activity level.
Primary Safety Endpoint | Time of surgery to 2 years post-surgery
  The primary safety endpoints listed below will be recorded as adverse events and qualified as to whether they are procedure or product related.
  • Adverse Events related to the procedure including:
  * Delayed wound healing (4wks post-surgery)
  * Wound infection (superficial or deep)
  * Neuritis (persistent 6wks post-surgery)
  * Peri-implant osteolysis
  * Reoperations of the index ankle
  * Revisions of the ligament repair Additionally, complications necessitating a return to OR due to implant failure, foreign body reaction, or deep wound infection will be captured and characterized.

SECONDARY OUTCOMES:
Physician Assessment of Healing | From 2 weeks post-surgery to 26 weeks post-surgery
  Subjects will complete post-surgery study follow-up visits during which time the physician assessment of healing will be completed.
Anterior Drawer Assessment | From 2 weeks post-surgery to 26 weeks post-surgery
  Subjects will complete post-surgery study follow-up visits during which time the anterior drawer assessment will be completed.
Talar Tilt Assessment | From 2 weeks post-surgery to 26 weeks post-surgery
  Subjects will complete post-surgery study follow-up visits during which time the talar tilt assessment will be completed.
Pain Medication Usage | From 2 weeks post-surgery to 26 weeks post-surgery
  Subjects will complete post-surgery study follow-up visits during which time the physician will document pain medication usage.
FAAM | From 2 weeks post-surgery to 26 weeks post-surgery
  The Foot and Ankle Ability Measure (FAAM) score is a percentage that indicates a patient's level of foot and ankle function. The FAAM is a survey that uses a 5-point Likert scale to score each item. The scale ranges from 4 for "no difficulty" to 0 for "unable to do". Patients can also select "not applicable" if the item doesn't apply to them.
FFI | From 2 weeks post-surgery to 26 weeks post-surgery
  The Foot Function Index (FFI) is a self-administered questionnaire that measures the impact of foot problems on a person's pain, disability, and activity restriction. The FFI uses a visual analog scale (VAS) to rate each item on a scale of 0 to 100, with higher scores indicating more pain, disability, or limitation.
CAIT | From 2 weeks post-surgery to 26 weeks post-surgery
  The Cumberland Ankle Instability Tool (CAIT) score is a number that indicates the severity of ankle instability. The CAIT score ranges from 0 to 30, with 30 being the best possible score and 0 being the worst.
VAS Pain | From 2 weeks post-surgery to 26 weeks post-surgery
  A VAS score is a measurement of pain intensity or other sensations and feelings using a visual analog scale. The VAS is scored by the following measures: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)
EQ-5D-5L | From 2 weeks post-surgery to 26 weeks post-surgery
  Consists of a 5-question measure where patients rate their health today on a 5-point scale on a 5-dimension scale and a visual analogue scale to measure overall health status.
Patient Satisfaction Scores | From 2 weeks post-surgery to 26 weeks post-surgery
  A subjective questionnaire measuring patient satisfaction will be collected follow-up visits.
FOTO | From 2 weeks post-surgery to 26 weeks post-surgery
  A subset of study sites will additionally collect FOTO data. The Focus on Therapeutic Outcomes (FOTO) is a numerical value that measures a patient's functional ability. Scores range from 0 (low function) to 100 (high function).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma & Extremities
Locations (8):
- United States (8):
  - MORE Foundation, Phoenix, Arizona
  - University of Florida, Gainesville, Florida
  - Southeast Orthopedic Specialists, Jacksonville, Florida
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Orthopedic Foot and Ankle Center, Worthington, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Health Houson, Houston, Texas
  - The Center for Advanced Orthopedics, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No
Unknown at this time.